CLINICAL TRIAL: NCT00006178
Title: Sirolimus Monotherapy to Optimize Activation Induced Cell Death (AICD) in Renal Transplants Following Lymphocyte Depletion Induction With Thymoglobulin
Brief Title: Sirolimus and Thymoglobulin to Prevent Kidney Transplant Rejection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000196; 00-DK-0196 (Other: NIDDK/NIH)
Record Dates: First submitted 2000-08-15; First posted 2000-08-16 (Estimated); Results first posted 2010-02-11 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2010-06

CONDITIONS: Kidney Failure
Keywords: Renal Failure; Anti-rejection; Apoptosis; Polyclonal Antibody; Kidney Transplant
MeSH Terms: conditions — Renal Insufficiency | interventions — Sirolimus; thymoglobulin

ARMS (1):
- Sirolimus and Thymoglobulin (Experimental): Thymoglobulin (Sangstat), a FDA-approved polyclonal rabbit-IgG antithymocyte preparation, will be given for ten days at the time of transplantation to achieve profound lymphocyte depletion. This will be paired with chronic therapy with Sirolimus (rapamycin, Wyeth-Ayerst), an oral immunosuppressant agent recently approved by the FDA.
  Interventions: Drug: Sirolimus; Drug: Thymoglobulin

INTERVENTIONS:
Drug: Sirolimus
Drug: Thymoglobulin

SUMMARY:
This study will test the safety and effectiveness of two drugs, Sirolimus and Thymoglobulin, for preventing rejection of transplanted kidneys. Standard anti-rejection therapy uses a combination of drugs, such as cyclosporine, tacrolimus, azathioprine, steroids, and others, that are taken daily for life. However, even with this daily therapy, more than half of kidney recipients slowly reject their transplant within 10 years. Both Thymoglobulin, an antibody, and Sirolimus, an anti-rejection drug, prevent rejection by lowering the response of the immune system to the transplanted organ. Thymoglobulin is given in the pre- and postoperative period, and Sirolimus is taken long term.

Patients who receive a kidney transplant at the National Institutes of Health Clinical Center are eligible for this study. Candidates will be screened with a medical history, physical examination, and blood and urine tests.

Participants will undergo a kidney transplant. Before the surgery, a central line (intravenous catheter), through which blood and medicine can be given, is placed in the neck or chest. Patients may also undergo leukapheresis, a procedure for collecting white blood cells. The cells can be stored for transfusion later if white cell counts drop following Thymoglobulin treatment. For this procedure, blood is drawn from a needle placed in the arm and flows into a machine that separates the blood components by spinning. The white cells are collected in a bag and the red cells and plasma are returned through a second needle in the other arm.

Thymoglobulin will be given intravenously the day before the transplant and days 1 through 9 after the operation. Sirolimus will be taken by mouth, mixed with water or orange juice. Sirolimus therapy starts the day of the transplant and continues for life.

Follow-up study visits will be scheduled weekly for the first month after the transplant, then every 6 months for 1 year and then once a year for 4 years. Procedures during these visits may include blood and urine tests, physical examination, and check of vital signs (i.e., blood pressure, heart rate, breathing rate, temperature). Kidney biopsies (removal of a small piece of tissue for examination under the microscope) will be done at 2 weeks, 1 month and 6 months after surgery and then yearly for 4 years to check for any damage to the kidney. In addition, a local doctor will do routine laboratory tests 2 to 3 times a week for the first 2 to 3 months aft...

DETAILED DESCRIPTION:
This protocol will test a novel dual agent combination therapy for its ability to prevent human renal allograft rejection. Thymoglobulin (Sangstat), a FDA-approved polyclonal rabbit-IgG antithymocyte preparation, will be given for ten days at the time of transplantation to achieve profound lymphocyte depletion. This will be paired with chronic therapy with Sirolimus (rapamycin, Wyeth-Ayerst), an oral immunosuppressant agent recently approved by the FDA. Rapamycin allows for antigen specific T cell activation but prevents T cell clonal expansion by interrupting IL-2 receptor beta-chain signal transduction. The rationale for this combination is to eliminate existing alloreactive T cell clones that could initiate a rejection at the time of transplantation, and to promote graft specific activation induced cell death (AICD) in repopulating T cells such that an allospecific T cell deficit is induced. The desired effect of this therapy is to prevent allograft rejection without the chronic use of calcineurin inhibitors or glucocorticosteroids, and in doing so, develop a regimen for transplantation that avoids most of the chronic drug toxicities inherent in the use of these two classes of immunosuppressants.

Twenty people will be evaluated in this pilot protocol. Ten will receive living donor kidney allografts and ten will receive cadaveric kidney allografts. Patients will be treated with Thymoglobulin beginning prior to graft implantation and continuing for ten days. Glucocorticosteroids will be given during the Thymoglobulin treatment to limit monocyte activation and prevent the cytokine release syndrome associated with this antibody preparation. Patients will be given Sirolimus orally beginning the day after transplantation and continuously thereafter. Patients will then be monitored for evidence of allograft rejection using standard functional parameters and protocol allograft biopsies. In addition, patients will be followed for a specific desired effect, allospecific AICD, that should promote the development of allospecific graft tolerance. This will be accomplished by assaying peripheral blood and allograft biopsies for apoptosis and peripheral blood for evidence of alloreactive T cell clone depletion.

ELIGIBILITY:
* INCLUSION CRITERIA:

Candidates for a kidney transplant performed at the NIH Clinical Center.

Willingness and legal ability to give informed consent.

Availability of donor tissue for testing. This could include splenic or peripheral blood lymphocytes from a cadaveric donor or a willing living donor enrolled on the Clinical Center Living Donor Protocol who consents to periodic phlebotomy for peripheral blood lymphocyte isolation.

EXCLUSION CRITERIA:

Immunosuppressive drug therapy at the time of or 2 months prior to enrollment. Specifically, candidates may not be taking prednisone, cyclosporine, tacrolimus, azathioprine, mycophenolate mofetil, anti-lymphocyte agents, cyclophosphamide, methotrexate, or other agents whose therapeutic effect is immunosuppressive.

Any active malignancy or any history of a hematogenous malignancy or lymphoma. Patients with primary, cutaneous basal cell or squamous cell cancers may be enrolled providing the lesions are appropriately treated prior to transplant.

Significant coagulopathy or requirement for anticoagulation therapy that would contraindicate protocol allograft biopsies.

Platelet count less than 100,000/mm(3).

Any known immunodeficiency syndrome.

Any history of cardiac insufficiency, major vascular disease, symptomatic coronary artery disease.

Systemic or pulmonary edema.

Inability to be effectively dialyzed.

Any condition that would likely increase the risk of protocol participation or confound the interpretation of the data.

Any history of sensitization to rabbits or extensive exposure to rabbits.

Inability or unwillingness to comply with protocol monitoring and therapy, including, among others, a history of noncompliance, circumstances where compliance with protocol requirements is not feasible due to living conditions, travel restrictions, access to urgent medical services, or access to anti-rejection drugs after the research protocol is completed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2000-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Matas AJ, Gillingham KJ, Sutherland DE. Half-life and risk factors for kidney transplant outcome--importance of death with function. Transplantation. 1993 Apr;55(4):757-61. doi: 10.1097/00007890-199304000-00014. PMID 8475549
- [Background] Morris PJ. Renal transplantation: a quarter century of achievement. Semin Nephrol. 1997 May;17(3):188-95. PMID 9165648
- [Background] Swanson SJ, Hale DA, Mannon RB, Kleiner DE, Cendales LC, Chamberlain CE, Polly SM, Harlan DM, Kirk AD. Kidney transplantation with rabbit antithymocyte globulin induction and sirolimus monotherapy. Lancet. 2002 Nov 23;360(9346):1662-4. doi: 10.1016/S0140-6736(02)11606-0. PMID 12457792
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2000-DK-0196.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus and Thymoglobulin: Thymoglobulin (Sangstat) will be given for ten days at the time of transplantation to achieve profound lymphocyte depletion. This will be paired with chronic therapy with Sirolimus (rapamycin, Wyeth-Ayerst)
Period: Overall Study
Arm/Group | Sirolimus and Thymoglobulin
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus and Thymoglobulin
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Secondary Outcome: Glomerular Filtration Rate (Flow Rate of Filtered Fluid Through the Kidney)
Description: measure 6 months after intervention
Time Frame: 6 month after intervention
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Sirolimus and Thymoglobulin
Number analyzed (Participants) | 12
mL/min | 69.1 (17.4)

2. Primary Outcome: Serum Creatinine Concentration
Description: measures at 6 months after intervention
Time Frame: 6 months after intervention
Population: Analysis includes all participants in the study. Analysis was per protocol.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Sirolimus and Thymoglobulin
Number analyzed (Participants) | 12
umol/L | 112 (34)

3. Primary Outcome: Serum Creatinine Concentration
Description: measures at 12 months after intervention
Time Frame: 12 months after intervention
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Sirolimus and Thymoglobulin
Number analyzed (Participants) | 12
umol/L | 107 (25)

4. Secondary Outcome: Glomerular Filtration Rate (Flow Rate of Filtered Fluid Through the Kidney)
Description: measure at 12 months after intervention
Time Frame: 12 months after intervention
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Sirolimus and Thymoglobulin
Number analyzed (Participants) | 12
mL/min | 74.2 (21.3)

ADVERSE EVENTS:
Arm/Group | Sirolimus and Thymoglobulin
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus and Thymoglobulin (N=12)
Acute cellular rejection (Renal and urinary disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus and Thymoglobulin (N=12)
varicella zoster reactivation (General disorders) | 1 (1)
bacterial urnary tract infection (Renal and urinary disorders) | 2 (2) — bacterial urinary tract infection with infected polycystic kidneys and a pretransplantation neurogenic bladder
diabetic foot cellulitis (Metabolism and nutrition disorders) | 1 (1) — diabetic foot cellulitis 15 months after transplantation
hernia (General disorders) | 2 (2)
lymphocoele (Immune system disorders) | 1 (1) — lymphocoele needing transperitoneal drainage
postpolio motor neuropathy (General disorders) | 1 (1) — postpolio motor neuropathy 1 year after transplantation responsive to intravenous immunoglobulin
Sirolimus-side-effect (diarrhoea) (General disorders) | 3 (3)
Sirolimus-side-effect (mouth ulcers) (General disorders) | 8 (8)
Sirolimus-side-effect (arthralgias) (General disorders) | 2 (2)
Sirolimus-side-effect (hyperlipidaemia) (General disorders) | 10 (10)

LIMITATIONS AND CAVEATS:
Optimal dose of RATG remains to be determined. Whether other depleting agents are as effective as RATG is unclear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes